CLINICAL TRIAL: NCT03886844
Title: Prolacta Compare. Growth and Weight Gain in Extremely Low Birth Weight Infants Fed an Exclusively Human Milk Based Diet With Prolacta®
Brief Title: Growth and Weight Gain in ELBW Infants Fed an Exclusively Human Milk Based Diet With Prolacta®
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Associate Professor for Pediatrics, Medical University of Vienna
Other Study IDs: Prolacta
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Weight Gain; Human Milk; Preterm Infants; Extremely Low Birth Weight
Keywords: Infant weight gain; Human milk fortifier; Preterm infants; ELBW infants
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prolacta group: Infants, who received a human milk fortifier based on human milk (12/2015-11/2018), started with an enteral intake of 100 ml/kg until 32 weeks corrected for prematurity
  Interventions: Dietary Supplement: Human milk fortifier based on human milk (Prolacta)
- "Frauenmilch Supplement"=FMS group: Infants, who received a human milk fortifier based on bovine milk (05/2012-06/2015), started with an enteral intake of 100 ml/kg

INTERVENTIONS:
Dietary Supplement: Human milk fortifier based on human milk (Prolacta) — Intervention is started with an enteral intake of 100 ml/kg until 32 weeks corrected for prematurity, afterwards a human milk fortifier based on bovine milk is administered until estimated date of birth or 52 weeks corrected for prematurity (weight <10. percentile) according to ESPGHAN(=European Society for paediatric gastroenterology, hepatology and nutrition) guidelines
  Groups: Prolacta group

SUMMARY:
Preterm infants are susceptible to postnatal growth restriction. Breast milk is the recommended source of nutrition for preterm infants. As preterm infants have enhanced nutritional requirements, multicomponent fortifiers are added to breast milk in order to establish adequate growth.

Due to the various benefits of human milk feds to preterm infants, a human milk fortifier based on donor milk (Prolact+6 H2MF® Prolacta, City of Industry, California) has been developed. With this study, the investigators want to evaluate the effect of human milk fortification on weight gain in extremely low birth weight infants (ELBW, <1000g birth weight) in comparison to bovine fortification.

DETAILED DESCRIPTION:
Preterm infants are susceptible to postnatal growth restriction. Breast milk is the recommended source of nutrition for preterm infants. Many positive short-term health effects like prevention necrotizing enterocolitis , effects on gut development and immunological issues are associated with breast milk feedings.

The composition of breast milk usually meets the nutritional demands of term infants. As preterm infants have enhanced nutritional requirements, multicomponent fortifiers are added to breast milk in order to establish adequate growth and proper neurodevelopmental outcome.

Due to the various benefits of human milk feds to preterm infants, a human milk fortifier based on donor milk (Prolact+6 H2MF® Prolacta, City of Industry, California) has been developed. This human milk fortifier contains more energy and protein than bovine milk fortifiers. So far, accurate data on growth and weight gain under an exclusive diet with human milk and the human milk fortifier Prolact+6H2MF®are missing. With this study, the investigators want to evaluate the impact of a human milk based fortifier on weight gain in extremely low birth weight infants (ELBW, <1000g birth weight) in comparison to bovine milk based fortifier.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a birth weight <1000 g

Exclusion Criteria:

* Congenital heart disease
* Major congenital birth defects
* Major inborn error of metabolism

Ages: 1 Day to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ELBW infants (extremely low birth weight infants, <1000g birth weight)
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2015-12; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
growth velocity g/kg/d at 37+0 weeks | at 37+0 weeks of gestation
  weight gain in g/kg/d

SECONDARY OUTCOMES:
growth velocity g/kg/d at 32+0 weeks | at 32+0 weeks of gestation
  weight gain in g/kg/d
growth velocity g/kg/d from start of fortification to 32+0 weeks | at 32+0 weeks of gestation
  weight gain in g/kg/d
Weight at 32+0 | at 32 weeks of gestation
  weight in grams
Weight at 37+0 | at 37+0 weeks of gestation
  weight in grams
Length at 32+0 | at 32+0 weeks of gestation
  Length in cm
Length gain at 32+0 | at 32+0 weeks of gestation
  Length gain in cm/week
Head circumference at 32+0 | at 32+0 weeks of gestation
  head circumference in cm
Head circumference gain at 32+0 | at 32+0 weeks of gestation
  head circumference gain in cm/week
Length at 37+0 | at 37 weeks of gestation
  Length in cm
Lengthgain at 37+0 | at 37 weeks of gestation
  Lengthgain in cm/week
Head circumference at 37+0 | at 37 weeks of gestation
  Head circumference in cm
Head circumference gain at 37+0 | at 37 weeks of gestation
  Head circumference gain in cm/week
Time to full enteral feeds | up to 37 weeks of gestation
  Day of life when full enteral feeds (140ml/kg) are tolerated
Incidence of necrotising enterocolitis | up to 37 weeks of gestation
  Necrotizing enterocolitis stage 2a according to Bell
Body composition | up to 6 months corrected for prematurity
  Fat and Fat- free mass measured by Body plethysmography
Blood parameter total protein | up to 37 weeks of gestation
  laboratory parameter
Blood parameter Urea | up to 37 weeks of gestation
  laboratory parameter
Blood parameter Triglyceride | up to 37 weeks of gestation
  laboratory parameter
Blood parameter Glucose | up to 37 weeks of gestation
  laboratory parameter
z- scores | at 37 weeks of gestation
  z-scores for weight , length and head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. PD. Nadja Haiden, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Paracelsus Medical University, Salzburg
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No